CLINICAL TRIAL: NCT04891822
Title: Enhanced Recovery After Bariatric Surgery(ERAS) in the Morbidly Obese Using Evidence-Based Clinical Pathways: A Prospective Observational Non-randomized Comparative Study
Brief Title: ERAS After Bariatric Surgery in Morbidly Obese
Status: Completed | Type: Observational
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, BON WOOK KOO, assistnat professor, Seoul National University Bundang Hospital
Other Study IDs: SNU-SLEEVE
Record Dates: First submitted 2021-04-23; First posted 2021-05-18 (Actual); Last update posted 2024-01-16 (Actual); Status verified 2024-01

CONDITIONS: ERAS; Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- E (ERAS protocol): receive ERAS protocol 8 hours of fasting and ingestion of oral carbohydrate 2 hour before surgery TIVA(Total intra-venous anesthesia) TAP(transversus abdominis plane) block IV-PCA using NSAIDs after surgery Resuming oral intake 2 hours after surgery.
  Interventions: Procedure: ERAS protocol
- C (Control): receive standard perioperative care 8 hours of fasting before surgery Inhalation anesthesia IV-PCA using NSAIDs Resuming oral intake 6 hours after surgery.

INTERVENTIONS:
Procedure: ERAS protocol — E: ERAS protocol C: control
  Groups: E (ERAS protocol)

SUMMARY:
Recently, the number of bariatric surgery is increasing but ERAS (Enhanced Recovery After Surgery) protocol for bariatric surgery needs revision with evidence. So we investigated usefulness of ERAS protocol for bariatric surgery in morbidly obese patients.

DETAILED DESCRIPTION:
Patients undergoing elective laparoscopic bariatric surgery are going to be recruited and divided into 2 groups: Group E will receive ERAS protocol, and Group C will receive standard perioperative care.

ERAS protocol comprises 8 hours of fasting and ingestion of oral carbohydrate 2 hour before surgery, TIVA(Total intra-venous anesthesia), TAP(transversus abdominis plane) block and IV-PCA using NSAIDs after surgery, and resumption of oral intake 2 hour after surgery.

Conventional anesthesia is composed of 8 hours of fasting, inhalation anesthesia, IV-PCA using NSAIDs, and resumption oral intake 6 hour after surgery.

In both groups, gastric ultrasonography will be used to measure gastric volume before surgery.

Functional hospital stay will be recorded from the end of surgery until all discharge criteria had been met. Pain scores will be recorded at 30 minutes, 4 hours, and 24 hours after surgery. Also, nausea and vomiting, time to ambulation, will be documented. After the patients are discharged, their charts are going to be reviewed and their medical expenses will be documented.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists grade 1 ~ 3
* BMI(Body Mass Index) ≥30
* Scheduled for elective laparoscopic bariatric surgery

Exclusion Criteria:

* American Society of Anesthesiologists grade 4 or 5
* History of abdominal surgery

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Morbidly obese patients undergoing elective laparoscopic bariatric surgery at Seoul National Bundang Hospital
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2021-06-02 (Actual); Primary Completion 2022-02-24 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Functional hospital stay | from end of surgery, until all discharge criteria had been met (an average of 3 days)
  time from the end of surgery until all discharge criteria had been met

SECONDARY OUTCOMES:
Postoperative Pain score | 30 minutes, 4 hours, and 24 hours after end of surgery
  100 mm scale of visual analogue scale (0~100mm)
Rescue drug and dosage | 30 minutes, 4 hours, and 24 hours after end of surgery
  Rescue drug and dosage for additional analgesia
Postoperative nausea and vomiting | until patient discharge (an average of 3 days)
  The presence or absence of postoperative nausea and vomiting
Time to ambulation | Time to ambulation (an average of 1 day)
  Time to ambulation after surgery
Medical expenses | until patient discharge (an average of 4 days)
  Medical expenses during inpatient (Korean won)

CONTACTS AND LOCATIONS:
Overall Officials: Bon Wook Koo, MD, Study Director — SNUBH
Locations (1):
- Seoul National Universuty, Bundang Hospital, Seongnam-si, Gyonggido, South Korea